CLINICAL TRIAL: NCT01284647
Title: A Prospective, Randomized, Double-blind, Double-dummy, Sucralfate Controlled, Multicenter Study to Evaluate the Efficacy of Teprenone On Chinese Patients With Chronic Non-Atrophic Erosive Gastritis
Brief Title: A Study to Evaluate the Efficacy of Teprenone On Chinese Patients With Chronic Non-Atrophic Erosive Gastritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Eisai China Inc. (Industry)
Responsible Party: Principal Investigator, Yinchun Zhang, Dr., Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-081
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Erosive Gastritis
Keywords: Chronic Erosive Gastritis; Teprenone; Sucralfate
MeSH Terms: interventions — geranylgeranylacetone; Sucralfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teprenone capsule (Experimental)
  Interventions: Drug: Teprenone capsule and placebo of sucralfate
- sucralfate (Active Comparator)
  Interventions: Drug: Sucralfate and placebo of teprenone

INTERVENTIONS:
Drug: Teprenone capsule and placebo of sucralfate — Teprenone 1 capsule (50mg)+placebo of sucralfate 4tab, tid×8 weeks.
  Arms: Teprenone capsule
Drug: Sucralfate and placebo of teprenone — Placebo of teprenone 1 capsule+ sucralfate 4 tab(1.0), tid×8 weeks
  Arms: sucralfate

SUMMARY:
The purpose of this study is to evaluate the efficacy of teprenone on chronic non-atrophic erosive gastritis and its therapeutic mechanism

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old
2. Have been diagnosed as chronic non-atrophic erosive gastritis by endoscopy within 1 weeks before enrollment, and the modified Lanza score ≥ 2
3. Have at least two symptoms in four major symptoms (epigastric pain, epigastric burning, early satiety, belching) and total symptom score ≥ 4 (Rome Ⅲ for Functional Gastrointestinal Disorders)

Exclusion Criteria:

1. Suspected upper gastrointestinal malignancy by endoscopy
2. Peptic ulcer and bleeding by endoscopy
3. Severe cardiac, hepatic or renal insufficiency
4. Severe neurological or psychological disease
5. Pregnant or lactating women
6. Have taken drugs which may affect evaluating the efficacy of study drug within two weeks before enrollment (includes but not limits to: Proton pump inhibitors such as omeprazole, rabeprazole, pantoprazole, lansoprazole, esomeprazole, H2 receptor antagonists such as cimetidine, ranitidine, famotidine, antacids such as calcium carbonate, gastric mucosal protectants such as colloidal bismuth potassium citrate and other bismuth products, sucralfate, aluminum phosphate, teprenone, gefarnate, aluminum magnesium carbonate, glutamine, rebamipide, ecabet, misoprostol, antibiotics such as amoxicillin, clarithromycin, tetracycline, ofloxacin, levofloxacin, furazolidone, metronidazole, tinidazole, Non-Steroid Anti-Inflammatory Drugs such as aspirin, ibuprofen, loxoprofen, naproxen, diclofenac, indomethacin, meloxicam, acetaminophen)
7. History of allergic reaction to the medications used in this study
8. Patients that investigators consider ineligible for this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The difference of the modified Lanza score after 4 weeks of treatment between teprenone group and sucralfate group | 0,4 weeks

SECONDARY OUTCOMES:
The difference of total effective rate after 4 weeks treatment evaluated by histologic examination on inflammation improvement between teprenone group and sucralfate group | 4 weeks
The difference of patients' gastric mucosal concentration of hexosamine, PGE2 and HSP70 after 4 weeks treatment between teprenone group and sucralfate group | 4 weeks
The difference of total effective rate after 4 and 8 weeks treatment evaluated by clinical symptom score between teprenone group and sucralfate group | 4 and 8 weeks
The difference of total effective rate after 8 weeks treatment evaluated by endoscopy between teprenone group and sucralfate group | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Principal Investigator — Changhai Hospital
Locations (8):
- China (8):
  - Tongren Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital of Xiamen University, Xiamen, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai Xinhua Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality